CLINICAL TRIAL: NCT02740075
Title: Effect of Mode of Transport Ventilation on Respiratory Parameters After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Edward O'Brien, Clinical Chief of Critical Care, University of California, San Diego
Other Study IDs: IRB# 150836
Record Dates: First submitted 2016-02-05; First posted 2016-04-15 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Complication of Ventilation Therapy
Keywords: Mechanical versus hand ventilation; Transport ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hand-ventilated: This group will be transported from the operating room to the intensive care unit with the anesthesia provider ventilating the patient by hand via Mapleson circuit and supplemental oxygen. Vital signs and end-tidal carbon dioxide will be monitored and recorded by one of the investigators. The anesthesia provider will be blinded to the end-tidal carbon dioxide levels and respiratory rate.
- Mechanically ventilated: This group will be transported from the operating room to the intensive care unit with the patient being ventilated by a transport ventilator with controlled tidal volume, respiratory rate, and positive end-expiratory pressure. Vital signs and end-tidal carbon dioxide will be monitored and recorded by one of the investigators.

SUMMARY:
After cardiac surgery patients are transported from the operating room (OR) to the intensive care unit (ICU) while intubated. Two principal methods of oxygenation and ventilation are used: (1) a transport ventilator or (2) a Mapleson Bag-Mask hand ventilating circuit. The choice of method is largely determined by the preference of the the anesthesiologist who is transporting the patient. The investigators postulate that the choice of either method might alter respiratory and hemodynamic parameters felt to be important for the immediate management of post-cardiac surgery patients. The investigators will prospectively record end-tidal carbon dioxide (ETCO2) (primary end-point) and change in minute volume, heart rate (HR), Blood pressure (BP), pulmonary artery (PA) pressures and cardiac output during transportation and upon arrival in the ICU. All of these variables are measured routinely but are not recorded. The investigators will compare patients transported with a ventilator to patients transported with a Mapleson circuit.

DETAILED DESCRIPTION:
After cardiac surgery, patients can have poor respiratory function and hemodynamics. The exact cause and contributing factors of this deterioration are not usually known and, often these patients demonstrate normal parameters at the end of surgery, but are significantly altered upon arrival in the ICU. Transportation of patients from the OR to the ICU is a period of significantly less intense monitoring and less well-controlled interventions (for example tidal volume (Vt) is largely arbitrary). Recent evidence suggests that the risk of intra-hospital transportation is significantly higher for ventilated patients than for all other patients. Some of this risk might be mitigated by the mode of ventilation because pulmonary and hemodynamic parameters are rarely measured during transportation. If the method used for ventilation and oxygenation during transport is important in maintaining stability upon presentation to the ICU, clinicians might choose one method over another. This would change clinical practice.

This is a prospective observational study assessing the effect of different modes of transport ventilation on respiratory and hemodynamic parameters on post cardiothoracic (CT) surgery patients admitted to the ICU. It is standard of care to measure peripheral blood CO2 (either end-tidal or arterial), minute volume, heart rate, blood pressure, cardiac output and pulmonary artery pressure for all patients admitted to the ICU after cardiac surgery. The investigators will simply record these values during transport and immediately on arrival in the ICU. At a 2 sided significance level of 0.05, the investigators will enroll 32 patients to detect a minimal difference from baseline ETCO2 of 15% at a power of 0.8.

The investigators will review each subjects medical record to obtain vital sign information and ventilatory parameters. The investigators will obtain individual HIPAA authorization from each subject.

All subjects will have just undergone cardiac surgery are intubated and are being transported to the ICU with either method of ventilation. The patients will be adult (age 18 and over who are competent to give their own consent). They will be recruited prior to surgery according to the inclusion and exclusion criteria listed below. No consideration will be made to gender, race, sexual orientation or national origin.

ELIGIBILITY:
Inclusion Criteria:

* Adults scheduled for elective cardiac surgery.
* No known pulmonary disease prior to surgery.

Exclusion Criteria:

* Patients who refuse to participate, patients under the age of 18, groups with known cognitive impairment, patients who are unable to consent or institutionalized individuals.
* Patients who are not expected to remain intubated after cardiac surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects will have just undergone cardiac surgery, are intubated, and are being transported to the ICU with either method of ventilation. Prospective research subjects will be identified from the list of patients scheduled for surgery on any given day. This list is published daily on a screen outside of the pre-operative area which is accessible to the public. Identifying prospective research subjects will not require access to medical record or review of private information.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Measure the collective differences in end-tidal carbon dioxide upon arrival in the ICU between mechanical ventilation and hand-ventilation | Baseline
Measure the collective differences in pulmonary arterial pressures upon arrival in the ICU between mechanical ventilation and hand-ventilation | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Edward O'Brien, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Thornton Hopsital, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schwebel C, Clec'h C, Magne S, Minet C, Garrouste-Orgeas M, Bonadona A, Dumenil AS, Jamali S, Kallel H, Goldgran-Toledano D, Marcotte G, Azoulay E, Darmon M, Ruckly S, Souweine B, Timsit JF; OUTCOMEREA Study Group. Safety of intrahospital transport in ventilated critically ill patients: a multicenter cohort study*. Crit Care Med. 2013 Aug;41(8):1919-28. doi: 10.1097/CCM.0b013e31828a3bbd. PMID 23863225
- [Background] Gillman L, Leslie G, Williams T, Fawcett K, Bell R, McGibbon V. Adverse events experienced while transferring the critically ill patient from the emergency department to the intensive care unit. Emerg Med J. 2006 Nov;23(11):858-61. doi: 10.1136/emj.2006.037697. PMID 17057138
- [Background] Warren J, Fromm RE Jr, Orr RA, Rotello LC, Horst HM; American College of Critical Care Medicine. Guidelines for the inter- and intrahospital transport of critically ill patients. Crit Care Med. 2004 Jan;32(1):256-62. doi: 10.1097/01.CCM.0000104917.39204.0A. PMID 14707589